CLINICAL TRIAL: NCT03812796
Title: Epigenetic Modulation of the immunE Response in GastrointEstinal Cancers (EMERGE)
Acronym: EMERGE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: 4SC AG (Industry); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR 4745
Record Dates: First submitted 2018-04-09; First posted 2019-01-23 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Cancer; GI Cancer
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms | interventions — domatinostat; avelumab

STUDY DESIGN:
Intervention Model Description: Non-randomised
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Domatinostat plus Avelumab (Experimental): This is a multicentre open-label, phase II non-randomised clinical trial domatinostat plus avelumab (two separate cohorts in phase IIB part of trial).
  Interventions: Drug: Domatinostat; Drug: Avelumab

INTERVENTIONS:
Drug: Domatinostat — Domatinostat is an oral tablet which will be given at a variable dose during the Phase IIA safety run in phase of the trial.
  During the Phase IIB efficacy phase of the trial patients will be treated with domatinostat at the safe and tolerated combination dose identified during the Phase IIA safety run in phase.
  Other Names: 4SC-202
Drug: Avelumab — Avelumab is a monoclonal antibody which is given via an intravenous infusion at a dose of 10mg/kg every two weeks on the first day of a two week cycle. (Day 1 q 14d) from Cycle 2 onwards.

SUMMARY:
A multicenter phase II non-randomised trial assessing the efficacy of domatinostat (4SC-202) plus avelumab in patients with GI cancer

DETAILED DESCRIPTION:
During this phase II non randomised trial patients with microsatellite stable colorectal or gastroesophageal cancer which has previously been treated with chemotherapy will be treated with domatinostat plus avelumab.

ELIGIBILITY:
Inclusion Criteria

i. Male/female patients aged ≥18 years ii. Histologically confirmed gastric, gastro-oesophageal junction or oesophageal adenocarcinoma (referred to as oesophagogastric adenocarcinoma (OGA) in this protocol) or colorectal adenocarcinoma (referred to as CRC in this protocol) iii. Agrees to undergo biopsies for translational endpoints iv. Tumour must be mismatch repair proficient assessed using a validated test such as immunohistochemistry for mismatch repair proteins or microsatellite instability testing v. Tumours should be advanced and inoperable or metastatic vi. Patients must have received at least one prior chemotherapy treatment for their cancer, have no established treatment option, or decides against an established treatment option.

vii. Adequate bone marrow function:

1. Absolute neutrophil count (ANC) ≥1.5 x109/L
2. White blood count >3x109/L
3. Platelets ≥100x109/L
4. Haemoglobin (Hb) ≥9g/dl (can be post-transfusion) viii. Adequate renal function: Creatinine Clearance o ≥30ml/min is required. This may be calculated as per local practice, if calculated CrCl is <60ml/min then EDTA is required to demonstrate CrCl of ≥30ml/min If available, the EDTA clearance should always take precedence over the creatinine clearance.

ix. Adequate liver function

a. Serum bilirubin ≤1.5x ULN b. ALT/AST ≤2.5x ULN or ALT/AST ≤5x ULN if metastatic disease to liver x. Adequate coagulation profile

1. International Normalised Ratio (INR) < 1.5
2. Activated Prothrombin Time (APTT) < 1.5xULN xi. Patients on oral anticoagulation are advised to change to low molecular weight heparin prior to study entry to be eligible xii. ECOG performance status 0-1 xiii. Patient is fit to undergo all protocol investigations and receive all protocol treatment based on the assessment oncology clinics xiv. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrolment.

xv. Willingness and ability to comply with the protocol for the duration of the study including scheduled visits, examinations, investigations and treatment plans xvi. Pregnancy must be excluded with a negative serum pregnancy test, within 7 days before initiation of therapy, if the risk of conception exists. Sexually active female patients must be surgically sterile or be postmenopausal or must agree to use highly effective contraception which must be used for 10 days before the negative pregnancy test. Sexually active male patients must be surgically sterile or must agree to use highly effective contraception, i.e. methods with a failure rate of <1% per year (see section 6.4 for full definition and examples of highly effective contraception). Highly effective contraception must be agreed to be used throughout the study and for 30 days after last avelumab treatment if risk of conception exists. Female patients of child-bearing potential should be strictly advised to use a highly effective contraceptive measure, from the time of screening to 30 days after the last dose of trial treatment. If the patient uses a hormonal contraceptive method, the patient's partner should additionally use a condom. Male patients with partners of child bearing potential should be strictly advised to use barrier contraception in addition to having their partner use another method of contraception during the trial and for three months after the last dose. Male patients should also be advised to abstain from sexual intercourse with pregnant or lactating women, or to use condoms.

Exclusion Criteria

i. Any contraindication or known hypersensitivity reaction to any of the study drugs ii. Persisting toxicity relating to prior therapy of >grade 1 CTCAE version 4.03 except alopecia of any grade and neuropathy ≤ grade 2, or other grade ≤2 not constituting a safety risk based on investigators judgement iii. Any prior treatment with immunotherapy including anti-PD-1or PD-L1 therapy or other immunomodulatory drugs.

iv. All subjects with brain metastases, except those meeting the following criteria:

1. Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrolment
2. No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
3. Subjects must be either off steroids or on a stable or decreasing dose of <10mg daily prednisone (or equivalent)

v. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 4.0), any history of anaphylaxis, or uncontrolled asthma (i.e., 3 or more features of partially controlled asthma) vi. Patients who have received chemotherapy or radiotherapy for a previous malignancy in the past 3 years.

vii. Any immunodeficiency disorder viii. Any active, known or suspected autoimmune disease that might deteriorate when receiving immunostimulatory agent, with the following exceptions:

1. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
2. Patients requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤10mg (or equivalent) of prednisolone per day
3. Administration of steroids through a route known to result in minimal systemic exposure (topical, intranasal, intra-ocular, intra-articular or inhalation) are acceptable. Steroids as pre-medication for hypersensitivity reactions e.g. CT contrast are also acceptable.

ix. Prior organ transplantation, including allogeneic stem-cell transplantation x. Active infection requiring systemic therapy xi. History of inflammatory bowel disease xii. Patients with a history of interstitial lung disease or radiological evidence of pulmonary fibrosis xiii. Cerebrovascular disease (including transient ischaemic attacks (TIA) and strokes) within the previous 6 months xiv. Cardiovascular diseases as follows:

1. Myocardial infarction within the previous 6 months
2. Unstable angina
3. Congestive heart failure ≥NYHA Classification Class II
4. Serious cardiac arrhythmia requiring medication (for example, ventricular tachycardia, supraventricular tachycardia or atrial fibrillation with a resting heart rate > 110bpm) xv. Current signs or symptoms of any other severe progressive or uncontrolled hepatic, haematologic, gastrointestinal, endocrine, respiratory or cardiac disease, which in the opinion of the investigator, might impair the subject's tolerance of trial treatment or procedures.

xvi. Major surgery, major trauma or open biopsy within 28 days prior to registration (not including staging laparoscopy) xvii. Evidence of bleeding diathesis or coagulopathy xviii. Active non-healing wound, ulcer or bone fracture requiring therapy xix. Known positive tests for human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome, hepatitis A or C virus, acute or chronic active hepatitis B infection xx. Use of live attenuated vaccine within 28 days of initiation of study therapy, or anticipation that a live attenuated vaccine will be required during the study xxi. Current lactation (patients that discontinue breastfeeding may be eligible) xxii. Other severe acute or chronic medical conditions or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety run-in phase: To establish a safe and tolerable dose of domatinostat in combination with avelumab for use in the main (Phase IIB efficacy) phase of the trial | The DLT period is 28 days following the first treatment with domatinostat and avelumab
  Progression through dosing levels will be determined by the occurrence of dose limiting toxicities in the study population.
Main Phase IIB (efficacy) phase: Objective response rate using RECIST 1.1 criteria | 6 months
  ORR defined as the proportion of patients with either CR or PR (assessed according to RECIST 1.1) by 6 months from combination treatment initiation. The best ORR will be presented as a proportion along side a 95% confidence interval

SECONDARY OUTCOMES:
Number of patients with adverse events (according to NCI-CTCAE version 4) as a measure of safety and tolerability | Up to 90 days after last dose
  Safety of domatinostat and avelumab will be assessed by summarizing adverse events as a proportion
Progression free survival according to RECIST 1.1 | upto 2 years
  PFS will be summarized using Kaplan Meier methods, presenting median survival with 95% confidence intervals. PFS is defined as the time from day of first treatment to disease progression or death from any cause. Patients without an event will be censored on day of last radiological follow up
Overall survival | upto 2 years
  OS will be summarized using Kaplan Meier methods, presenting median survival with 95% confidence intervals. OS is defined as the time from say of first treatment to death from any cause. Alive patients will be censored at the last follow up date
Disease control rate | At 6 and 12 months on treatment
  The proportion of patients with best disease control (CR, PR or SD) at 6 months and 12 months from initiation of combination treatment will be presented with a 95% confidence interval
Duration of objective response according to RECIST 1.1 | upto 2 years
  DoOR will be summarized using Kaplan Meier methods. DoOR is defined as the time between the initial response to treatment and subsequent disease progression or relapse. Patients without an event will be censored on day of last radiological assessment

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Consultant Medical Oncologist
Locations (2):
- United Kingdom (2):
  - The Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey
  - The Royal Marsden Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cartwright E, Slater S, Saffery C, Tran A, Turkes F, Smith G, Aresu M, Kohoutova D, Terlizzo M, Zhitkov O, Rana I, Johnston EW, Sanna I, Smyth E, Mansoor W, Fribbens C, Rao S, Chau I, Starling N, Cunningham D. Phase II trial of domatinostat (4SC-202) in combination with avelumab in patients with previously treated advanced mismatch repair proficient oesophagogastric and colorectal adenocarcinoma: EMERGE. ESMO Open. 2024 Apr;9(4):102971. doi: 10.1016/j.esmoop.2024.102971. Epub 2024 Mar 21. PMID 38518549